CLINICAL TRIAL: NCT03920748
Title: Evaluation of the Relationship Between Airway Measurements With Ultrasonography and Laryngoscopic View in Newborn and Infants
Brief Title: Evaluation of the Relationship Between Airway Measurements and Laryngoscopic View in Newborn and Infants
Status: Completed | Type: Observational
Sponsor: Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Feyza Sever, Specialist physician, Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital
Other Study IDs: 2018105
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia Intubation Complication; Infant; Newborn
Keywords: Difficult laryngoscopy, airway measurements, newborn, infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult laryngoscopy (Group D): Glottic structures appearing during laryngoscopy are graded according to Cormack-Lehane (CL) Classification. According to this classification, patients are divided into two groups, patients with grade 3-4 are classified as difficult laryngoscopy ( Group D).
  Interventions: Other: Group D
- Easy laryngoscopy (Group E): Glottic structures appearing during laryngoscopy are graded according to Cormack-Lehane (CL) Classification. According to this classification, patients are divided into two groups, patients with grade 1-2 are classified as easy laryngoscopy ( Group E).
  Interventions: Other: Group E

INTERVENTIONS:
Other: Group D — According to Cormack-Lehane (CL) Classification; laryngoscopic view grade 3-4 is defined as Group D
  Groups: Difficult laryngoscopy (Group D)
Other: Group E — According to Cormack-Lehane (CL) Classification; laryngoscopic view grade 1-2 is defined as Group E
  Groups: Easy laryngoscopy (Group E)

SUMMARY:
Background and Aim: The overall incidence of difficult laryngoscopy in pediatric anesthesia is lower than in adults, but this risk is higher in patients younger than one year of age. In the last decade, different measurements have been used to obtain difficult laryngoscopy markers in children. In this study, we aimed to evaluate the relationship between the airway measurements (some performed by using ultrasonography (USG)) and the difficult laryngoscopic view in neonates and infants.

Design: This is a prospective, single blinded, observational study. The number of patients was calculated as follows: A sample of 12 from the positive group (difficult laryngoscopy group) and 96 from the negative group (easy laryngoscopy group) achieve 80% power to detect a difference of 0.25 between the area under the ROC curve (AUC) under the null hypothesis of 0.50 and an AUC under the alternative hypothesis of 0,75 using a two-sided z-test at a significance level of 0.05.

Methods: All patients which is newborn and infant age group undergoing elective surgery requiring intubation under general anesthesia are assessed. Patients' age, body mass index (BMI), thyromental distance, mandibula length, the distance between the lip corner and ipsilateral ear tragus, and the transverse length (measured by hand sign-middle-ring fingers adjacent side by side) measurements are recorded. In thyromental distance measurement, "thyroid notch" are determined by USG.

The laryngoscopic view is graded by a different experienced anaesthetist who is blinded to the airway measurements.

Statistical analysis:

Receiver operating characteristic (ROC) curves are used to determine the best cut-off point for distance variables in the separation of difficult and easy laryngoscopy groups. Sensitivity, selectivity, positive predictive value and negative predictive values of lengths are calculated according to determined cut point.The difference between the two groups in terms of qualitative variables are evaluated by chi-square or Fisher's exact test. The normal distribution of the numerical variables are examined with the Shapiro-Wilk test. The difference between the two groups in terms of numerical variables are investigated by Mann Whitney U test. Values of p <0.05 are considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Newborn and infant age group
* Undergoing elective surgery requiring intubation under general anesthesia

Exclusion Criteria:

* History of congenital maxillofacial defect,
* History of upper airway pathology (tumor, cleft palate-lips, etc.)
* History of head and neck trauma (fracture, swelling, scar )

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn and infant age group undergoing elective surgery at Ankara Childrens' Health and Diseases Hematology Oncology Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Thyromental distance (TMD) | 1 hour
  The thyromental distance, unit of measure cm, is detected using a US linear probe with the transducer placed in the transverse plane. Thyromental distance is measured in cm as straight line from thyroid notch to lower border of mentum with head extended in all patients.
Other airway measurements | 1 hour
  The other primary objective of this study is to identify if any preanesthetic airway assessment maneuvers (such as mandibula length, the distance between the lip corner and ipsilateral ear tragus, and the transverse length (measured by hand sign-middle-ring fingers adjacent side by side) measurements) would be associated with difficult laryngoscopy in newborn and infants.

SECONDARY OUTCOMES:
Demographic data | 1 hour
  The secondary objective of this study is to identify if factors such as age, sex, bady mass index (BMI) and physical status grade would be associated with grade III and IV laryngoscope views in newborn and infants.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sever, Principal Investigator — Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital
Locations (1):
- Ankara Childrens' Health and Diseases Hematology Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)